CLINICAL TRIAL: NCT05699616
Title: Laparoscopic Management of Perforated Peptic Ulcer: Multicenter Experience
Brief Title: Management of Perforated Peptic Ulcer
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Abdallah Mohamed Taha Aly, Assistant Professor, South Valley University
Other Study IDs: SVU-MED-SUR011-4-22-10-466
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Perforated Peptic Ulcer
Keywords: Peptic ulcer; Laparoscopic repair; Open repair; Graham Patch
MeSH Terms: conditions — Peptic Ulcer Perforation; Peptic Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Repair of perforated peptic ulcer — Repair of perforated peptic ulcer either open or laparoscopic.

SUMMARY:
Perforated peptic ulcer (PPU) is a common surgical emergency. Exploratory laparotomy and repair with the omental patch are routine surgical intervention till now. In developing counties, laparoscopic repair is still not considered the gold standard in this emergency condition. This study was conducted to evaluate laparoscopic management of PPU in terms of peri-operative outcomes.

DETAILED DESCRIPTION:
Files of all patients admitted to our hospital with perforated peptic ulcer in the last 4 years and underwent operative management.

Demographic, clinical and perioperative outcomes will be collected tabulated and analyzed.

ELIGIBILITY:
Inclusion Criteria:

- All patients with perforated peptic ulcer admitted to our hospital in last 4 years and underwent surgical intervention.

Exclusion Criteria:

Uncompleted patents files.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with perforated peptic ulcer admitted to our hospital in last 4 years and underwent surgical intervention.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Operative time | 2 hours
  Time from skin incision to skin closure
Leakage | 5 days
  Leakage from the repair
Time to return to normal daily activities. | 2 weeks
  Time to return to normal daily activities after surgery.
Perioperative complications | 1 month
  Any encountered perioperative complications related to surgical intervention..

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah M Taha, MD, Principal Investigator — South Valley University
Locations (1):
- Qena Faculty of Medicine, South Valley University Hospitals, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bertleff MJ, Halm JA, Bemelman WA, van der Ham AC, van der Harst E, Oei HI, Smulders JF, Steyerberg EW, Lange JF. Randomized clinical trial of laparoscopic versus open repair of the perforated peptic ulcer: the LAMA Trial. World J Surg. 2009 Jul;33(7):1368-73. doi: 10.1007/s00268-009-0054-y. PMID 19430829
- [Background] Lunevicius R, Morkevicius M. Management strategies, early results, benefits, and risk factors of laparoscopic repair of perforated peptic ulcer. World J Surg. 2005 Oct;29(10):1299-310. doi: 10.1007/s00268-005-7705-4. PMID 16132404
- [Background] Katkhouda N, Mavor E, Mason RJ, Campos GM, Soroushyari A, Berne TV. Laparoscopic repair of perforated duodenal ulcers: outcome and efficacy in 30 consecutive patients. Arch Surg. 1999 Aug;134(8):845-8; discussion 849-50. doi: 10.1001/archsurg.134.8.845. PMID 10443807
- [Background] Lagoo S, McMahon RL, Kakihara M, Pappas TN, Eubanks S. The sixth decision regarding perforated duodenal ulcer. JSLS. 2002 Oct-Dec;6(4):359-68. PMID 12500837
- [Background] Quah GS, Eslick GD, Cox MR. Laparoscopic Repair for Perforated Peptic Ulcer Disease Has Better Outcomes Than Open Repair. J Gastrointest Surg. 2019 Mar;23(3):618-625. doi: 10.1007/s11605-018-4047-8. Epub 2018 Nov 21. PMID 30465190